CLINICAL TRIAL: NCT05902260
Title: The Effects of an Oncology Tailored Nutritional Intervention on the Bioavailability and Immune-activity of PD-1 Immune Checkpoint Inhibitors in Patients with Lung Cancer
Brief Title: The Effects of an Nutritional Intervention on PD-1 ICI in NSCLC
Acronym: NutriCim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joachim Aerts, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Joachim Aerts, MD PhD, Prof dr, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC2021-0104
Record Dates: First submitted 2023-03-07; First posted 2023-06-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: immunotherapy; nutritional intervention
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutritional intervention (Experimental): Subjects should consume two 200 mL bottles of study product per day
  Interventions: Dietary Supplement: Nutritional intervention; Drug: Immunotherapy

INTERVENTIONS:
Dietary Supplement: Nutritional intervention — Subjects should consume two 200 mL bottles of study product per day next to their cancer treatment (immunotherapy)
Drug: Immunotherapy — Pembrolizumab monotherapy with or without combination chemotherapy according to standard of care

SUMMARY:
Over 65% of all lung cancer patients experience significant weight loss fuelled by a catabolic state that is represented by enhanced protein breakdown. The metabolic state of patients is a key effector of protein clearance, and the increased albumin as well as monoclonal antibodies clearance that is observed in patients with progressive cancer disease inversely correlates with treatment response and may well be consequential to changes in the metabolic state of cancer patients. Interestingly, several studies in cancer patients receiving chemotherapy, amongst which are NSCLC patients, have shown that weight loss and catabolism can be prevented or improved by intake of high energy/high protein Oral Nutritional Supplements (ONS). An increased clearance of anti-PD-1 ICI may also represent a general dysfunctioning of the immune system, because immune cell activation, proliferation, migration and tumor cell killing may all be influenced by cachexia. Enrichment of nutritional supplements with specific nutrients known to have immune-modulating properties, may further balance immune responses supportive of ICI efficacy.

The investigators hypothesize that high energy/high protein nutritional supplements decrease protein clearance including drug clearance in NSCLC patients receiving anti-PD-1 ICIs, which on its turn would positively affect anti-PD-1 drug bioavailability, leading to activation of the immune system and thereby an increased response to PD-1 ICIs.

The primary aim is to investigate the variability of clearance during a 12-weeks nutritional intervention period. The secondary aim is to investigate the feasibility for the subjects to comply with the study protocol. Lastly, the investigators aim to study the feasibility of gathering data on a number of exploratory parameters that may link nutritional intake to clinically relevant outcomes.

DETAILED DESCRIPTION:
Rationale: Over 65% of all lung cancer patients experience significant weight loss fuelled by a catabolic state that is represented by enhanced protein breakdown. The metabolic state of patients is a key effector of protein clearance, and the increased albumin as well as monoclonal antibodies clearance that is observed in patients with progressive cancer disease inversely correlates with treatment response and may well be consequential to changes in the metabolic state of cancer patients. Interestingly, several studies in cancer patients receiving chemotherapy, amongst which are NSCLC patients, have shown that weight loss and catabolism can be prevented or improved by intake of high energy/high protein Oral Nutritional Supplements (ONS).

The investigators hypothesize that high energy/high protein nutritional supplements decrease protein clearance including drug clearance in NSCLC patients receiving anti-PD-1 ICIs, which on its turn would positively affect anti-PD-1 drug bioavailability, leading to activation of the immune system and thereby an increased response to PD-1 ICIs.

An increased clearance of anti-PD-1 ICI may also represent a general dysfunctioning of the immune system, because immune cell activation, proliferation, migration and tumor cell killing may all be influenced by cachexia. Enrichment of nutritional supplements with specific nutrients known to have immune-modulating properties, may further balance immune responses supportive of ICI efficacy.

In conclusion, nutritional intervention with high energy/high protein nutritional supplements, especially if enriched with nutrients known for their immune- or microbiome-modulation properties, may have a positive impact on several mechanisms underlying cachexia-induced PD-1 ICI efficacy impairment.

Objective: The primary aim is to investigate the variability of clearance during a 12-weeks nutritional intervention period. The secondary aim is to investigate the feasibility for the subjects to comply with the study protocol. Lastly, the investigators aim to study the feasibility of gathering data on a number of exploratory parameters that may link nutritional intake to clinically relevant outcomes.

Study design: NutriCim is a feasibility study specifically designed to gather information on:

(i) the rate of NSCLC patient recruitment,(ii) the feasibility of collecting relevant data (compliance to protocol), and (iii) the effects of nutritional intervention on a number of parameters representing the patients' nutritional, immune, and microbiome status with a primary focus on pembrolizumab clearance.

Patients will start with the daily nutritional intervention prior to start of the first infusion of anti-PD-1 ICI immunotherapy and will continue this nutritional support for 4 treatment cycles, corresponding with 12 weeks of treatment. Blood samples, questionnaires and faecal specimens will be collected on several time points during this treatment. Changes from baseline for the different parameters on an individual patient level will, taking into account nutritional supplements compliance, be compared to patient outcomes, as well as with a historical cohort of NSCLC patients on similar treatment not receiving nutritional supplements.

ELIGIBILITY:
Inclusion criteria:

* Capable of oral intake and digestion of the nutritional test product
* Subjects with cytologically confirmed Stage IV or recurrent NSCLC, who have not received prior systemic therapy treatment for their advanced NSCLC. Completion of treatment with cytotoxic chemotherapy, biological therapy, and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as therapy was completed at least 6 months prior to the diagnosis of metastatic disease.
* Subjects must have programmed death-ligand 1 (PD -L1) immunohistochemical (IHC) testing.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Measurable disease by CT per response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) criteria
* Adequate haematological, renal and liver function

Exclusion criteria:

* Subject with an active auto-immune disease requiring systemic treatment
* Lung disease requiring systemic steroids in doses of >10 mg prednisolone (or equivalent dose of other steroid)
* Previous allogeneic or organ transplant Serious concomitant systemic disorders (for example active infection, unstable cardiovascular disease) which in the opinion of the investigator would compromise the patient's ability to complete the study, or would interfere with the evaluation of the efficacy and safety of the study treatment
* Known positive test for hepatitis B virus or hepatitis C virus or human immunodeficiency virus (HIV) indicating acute or chronic infection
* Allergy to cow's milk protein, soy or fish, requiring a fibre-free diet or suffering galactosemia or lactose intolerance
* Moderate to severe hypercalcemia, i.e. total calcium level corrected for albumin ≥14.0 mg/dL (3.5 mmol/L)
* Patient has had other malignancies within the past 3 years, except for stable non-melanoma skin cancer, fully treated and stable early stage prostate cancer or carcinoma in situ of the cervix or breast without need of treatment
* Simultaneous participation in other clinical trial
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
The variability of clearance of pembrolizumab during a 12-weeks nutritional intervention period in NSCLC patients receiving anti PDL-1 treatment, | from baseline to end of study (16 weeks)
  Blood for pharmacokinetic analysis and biomarker analysis will be withdrawn in a 5 mL serum tube

SECONDARY OUTCOMES:
Feasibility of recruiting 50 patients in 1.5 year for this study | 1.5 year after first inclusion
  Recruitment rate of patient inclusion, every patient eligible for this study will be asked for enrollment
Feasibility for the subjects to comply with the study protocol | from baseline to 16 weeks (end of study)
  Rate of compliance to the study procedures including the intake of the nutritional intervention and the feasibility of data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Aerts, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided